CLINICAL TRIAL: NCT05653752
Title: A Phase 1, Multicenter, Open-label, First-in-human Study of YL202 in Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer and Breast Cancer
Brief Title: A Study of YL202 in Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer and Breast Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: MediLink Therapeutics (Suzhou) Co., Ltd. (Industry)
Collaborators: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YL202-INT-101-01
Record Dates: First submitted 2022-12-01; First posted 2022-12-16 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Non Small Cell Lung Cancer; Breast Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- YL202 Dose escalation (Experimental): YL202 will be administrated intravenously (IV) per dose level in which the patients are assigned.
  Interventions: Drug: YL202

INTERVENTIONS:
Drug: YL202 — YL202 is provided as the lyophilized powder, 200 mg/vial. YL202 will be given intravenously once every 3 weeks (Q3W) as a cycle.
  The initial dose of YL202 will be infused IV into each patient for 90 ±10 minutes. If there is no infusion-related reaction after the initial dose, the second and subsequent doses of YL202 will be infused IV into each patient for 60 ±10 minutes.

SUMMARY:
This is a phase 1, multicenter, open-label, first-in-human study of YL202 conducted in the United States and China.

The study will evaluate the safety and tolerability of YL202 in patients with locally advanced or metastatic epidermal growth factor receptor (EGFR)-mutated NSCLC or hormone receptor (HR)-positive and HER2-negative BC, which have been heavily treated by standard treatment.

ELIGIBILITY:
Inclusion Criteria

Patients must satisfy all of the following criteria to be included in the study:

1. Informed of the trial before the start of the trial and voluntarily sign their name and date on the informed consent form
2. Aged ≥18 years
3. Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 to 2
4. Adequate organ and bone marrow function, defined as follows:

   * Hemoglobin ≥9.0 g/dL (have not received blood transfusion or erythropoietin treatment within 14 days before the first dose)
   * Absolute neutrophil count ≥1.5 × 109/L (have not received granulocyte colony-stimulating factor or granulocyte-macrophage colony-stimulating factor treatment within 14 days before the first dose)
   * Platelet count ≥100 × 109/L if no demonstrable hepatic metastases or ≥75 × 109/L in the presence of hepatic metastases (have not received platelet transfusion, thrombopoietin, or interleukin-11 treatment within 14 days before the first dose)
   * TBIL ≤1.5 × ULN if no demonstrable hepatic metastases or ≤3 × ULN in the presence of hepatic metastases
   * ALT and AST ≤3 × ULN if no demonstrable hepatic metastases or ≤5 × ULN in the presence of hepatic metastases
   * Serum albumin ≥2.5 g/dL
   * Creatinine clearance ≥60 mL/min (calculated according to Cockcroft Gault formula)
   * Activated partial thromboplastin time and international normalized ratio ≤1.5 × ULN, except for patients receiving anticoagulant therapy, who must have international normalized ratio within therapeutic range as deemed appropriate by the investigator
5. Female patients of childbearing potential must agree to use a highly effective form of contraception and not donate, or retrieve for their own use, ova from the time of screening and throughout the study period, and for at least 6 months after the last dose of study drug. Male patients must agree to use a highly effective form of contraception and not freeze or donate sperm from the time of screening and throughout the study period, and for at least 6 months after the last dose of study drug.
6. Life expectancy of ≥3 months
7. Able and willing to comply with protocol visits and procedures
8. For NSCLC patients:

   * Have a histologically or cytologically confirmed diagnosis of locally advanced or metastatic NSCLC not amenable to curative surgery or radiation
   * Have a documentation of an EGFR-activating mutation (exon 19 deletion or L858R) detected from tumor tissue at diagnosis or thereafter. Participants who have this EGFR mutation detected from blood sample may be eligible on a case-by-case basis after discussion with the sponsor.
   * Have documentation of disease progression on or after, or are intolerant to most recent treatment regimen for locally advanced or metastatic disease. Participants must have received all of the following:

     * Prior treatment with a regimen containing a 3rd-generation EGFR TKI (e.g., osimertinib). Patients receiving a 3rd-generation EGFR TKI at the time of signing informed consent should continue to take the EGFR TKI until 5 days prior to Cycle 1 Day 1
     * Systemic therapy with at least 1 platinum-based chemotherapy regimen
     * Participants in the US must have also received prior treatment with an anti-PD-(L)1 antibody, unless they have high-risk factors indicating preferable avoidance of anti-PD-(L)1 therapy (e.g., intolerance or lack of efficacy is anticipated) Note: Patients who received platinum-based chemotherapy concurrently with anti-PD-(L)1 antibody as one regimen are eligible.

   For BC patients:
   * Have a histologically or cytologically confirmed diagnosis of unresectable locally advanced or metastatic HR-positive and HER2-negative (IHC 0, 1+, 2+/ISH-) BC (per American Society of Clinical Oncology-College of American Pathologists [ASCO-CAP] guidelines)
   * Have documentation of disease progression on or after, or were intolerant to at least 1 prior line of endocrine therapy in combination with a CDK4/6 inhibitor
   * Have received 0-4 lines of chemotherapy regimens (including ADCs) for locally advanced or metastatic disease

   Note 1: Prior treatments with PI3K inhibitors, mTOR inhibitors, AKT inhibitors, and PARP inhibitors are allowed.

   Note 2: If a patient develops disease relapse/progression during or within 6 months after the end of the (neo-)adjuvant therapy, or radical radiotherapy and chemotherapy, the treatment regimen will be counted as one line of treatment for locally advanced or metastatic disease, for the purpose of this inclusion criteria.
9. Have at least 1 measurable tumor lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
10. Willing to provide archival or fresh tumor tissue samples for assessment of HER3 expression level. Patients who are not able to provide tumor samples or have inadequate samples may be eligible after discussion with the sponsor.

Exclusion Criteria

Patients who meet any of the following criteria will be disqualified from entering the study:

1. Prior treatment with an agent targeting HER3 (including antibody, ADC, chimeric antigen receptor T cell [CAR-T], and other drugs)
2. Intolerant to prior treatment with a topoisomerase I inhibitor or an ADC that consists of a topoisomerase I inhibitor, including but not limited to topotecan, irinotecan, and DXd (e.g., severe diarrhea)
3. Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
4. Inadequate washout period for prior anticancer treatment before the first dose of study drug, defined as follows:

   * Any cytotoxic chemotherapy or small molecular-targeted therapy (other than EGFR TKI) <2 weeks or 5 half-lives, whichever is shorter
   * Endocrine therapy <3 weeks
   * Monoclonal antibodies or other biological therapy <3 weeks
   * Herbal medicine with antitumor indications <2 weeks
   * Whole brain radiation therapy <2 weeks or stereotactic brain radiation therapy <1 week
   * Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation <4 weeks or palliative radiation therapy <2 weeks
5. Undergone major surgery (not including diagnostic surgery) within 4 weeks before the first dose of study drug or expect major surgery during the study
6. Prior allogeneic bone marrow transplantation or solid-organ transplantation
7. Received systemic steroids (>20 mg/day of prednisone or its equivalent) or other immunosuppressive therapy within 2 weeks before the first dose of study drug. The following are exceptions to this criterion:

   * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
   * Systemic steroids at physiological doses as replacement therapy (e.g., physiological corticosteroid replacement therapy for adrenal or pituitary insufficiency)
   * Steroids as premedication for hypersensitivity reactions (e.g., computed tomography [CT] scan premedication) or steroids as antiemetic premedication
8. Received any live vaccine within 4 weeks before the first dose of study drug or intend to receive a live vaccine during the study
9. A history of leptomeningeal carcinomatosis
10. Brain metastases or spinal cord compression unless asymptomatic or treated and stable off steroids and anti-convulsants for at least 2 weeks before the first dose of study drug
11. Uncontrolled or clinically significant cardiovascular disease, including but not limited to:

    * Medical history of symptomatic congestive heart failure (New York Heart Association class II to IV) or any arterial thromboembolic event (e.g., myocardial infarction, unstable angina, cerebrovascular accident, and transient ischemic attack) within 6 months before the first dose
    * Uncontrolled hypertension, defined as systolic blood pressure (SBP) >160 mm Hg and/or diastolic blood pressure (DBP) >100 mm Hg after antihypertensive therapy
    * Serious cardiac arrhythmia that requires treatment
    * Corrected QT interval by Fridericia's formula (QTcF) prolongation to >470 ms
12. A history of (noninfectious) interstitial lung disease (ILD)/pneumonitis that requires steroids, current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening
13. Clinically significant concomitant pulmonary disease, including but not limited to:

    * Pulmonary embolism within 3 months of the start of study treatment
    * Any autoimmune, connective tissue, or inflammatory disorder (e.g., rheumatoid arthritis, Sjögren's syndrome, sarcoidosis) where there is documented or suspicion of pulmonary involvement at the time of screening
    * Prior complete pneumonectomy
14. Patients with active or chronic corneal disorders, or patients with other active ocular conditions requiring ongoing therapy or with any clinically significant corneal disease that prevents adequate monitoring of drug-induced keratopathy.
15. Have a diagnosis of Gilbert's syndrome
16. Uncontrolled third-space fluid (e.g., pleural effusions, ascites, pericardial effusions) that requires repeated drainage
17. Active gastric and duodenal ulcers, ulcerative colitis, or other gastrointestinal conditions that may cause bleeding or perforation by the investigator's discretion
18. Active infection that requires systemic therapy within 1 week before the first dose. Patients receiving prophylactic anti-infective therapy (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) may be eligible after discussion with the sponsor.
19. Known human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV) infection. Patients with HIV, HBV, or HCV infection may be enrolled after evaluation of eligibility based on FDA's guideline Cancer Clinical Trial Eligibility Criteria: Patients with HIV, Hepatitis B Virus, or Hepatitis C Virus Infections
20. Any other primary malignancy within 3 years before the first dose of study drug, except adequately resected non-melanoma skin cancer, curatively treated in situ disease, or other curatively treated solid tumors
21. Unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia and pigmentation) not yet resolved to NCI CTCAE Grade ≤1, baseline, or the level specified in the inclusion/exclusion criteria. Patients with chronic Grade 2 toxicities who are asymptomatic or adequately managed with stable medication may be eligible after discussion with the sponsor.
22. A history of severe hypersensitivity reactions to the drug substances, inactive ingredients in the drug product, or other monoclonal antibodies
23. Women who are breastfeeding or pregnant as confirmed by pregnancy tests performed within 3 days before the first dose
24. Any illness, medical condition, organ system dysfunction, or social situation, including but not limited to mental illness or substance/alcohol abuse, deemed by the investigator to be likely to interfere with a patient's ability to sign informed consent, adversely affect the patient's ability to cooperate and participate in the study, or compromise the interpretation of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-12-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the occurrence of DLTs during the first cycle | At the end of Cycle 1 (each cycle is 21 days)
Evaluate the AEs as characterized by type, frequency, severity, timing, seriousness and relationship to study treatment | By the global end of trial date, approximately within 36 months

SECONDARY OUTCOMES:
Characterize the PK parameter AUC | Approximately within 36 months
Characterize the PK parameter Cmax | Approximately within 36 months
Characterize the PK parameter Ctrough | Approximately within 36 months
Characterize the PK parameter CL | Approximately within 36 months
Characterize the PK parameter Vd | Approximately within 36 months
Characterize the PK parameter t1/2 | Approximately within 36 months
Assess the incidence of anti-YL202 antibodies | Approximately within 36 months
Evaluate the objective response rate (ORR) | Approximately within 36 months
  ORR: defined as the proportion of patients who achieved a best overall response of complete response (CR) or partial response (PR).
Evaluate the disease control rate (DCR) | Approximately within 36 months
  DCR: defined as the proportion of patients who achieved a best overall response of CR, PR or stable disease (SD).
Evaluate the best tumor response | Approximately within 36 months
  Best tumor response: defined as the maximum percentage change in the sum of longest dimensions of measurable lesion(s) at any time during the study.

OTHER OUTCOMES:
Evaluate the duration of response (DoR) | Approximately within 36 months
  DoR: defined as the time interval from the date of the first documentation of objective response (CR or PR) to the date of the first documentation of PD. The DoR will be assessed for patients with a response (CR or PR) only.
Evaluate the time to response (TTR) | Approximately within 36 months
  TTR: defined as the time interval from the date of the first dose of study drug to the date of the first documentation of objective response (CR or PR).
Evaluate the progression-free survival (PFS) | Approximately within 36 months
  PFS: defined as the time interval from the date of the first dose of study drug to the date of first documentation of PD or death due to any cause, whichever occurs first.
Evaluate the overall survival (OS) | Approximately within 36 months
  OS: defined as the time interval from the date of the first dose of study drug to the date of death due to any cause.

CONTACTS AND LOCATIONS:
Locations (13):
- United States (7):
  - BRCR Global, Plantation, Florida
  - Karmanos Cancer Institute, Detroit, Michigan
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Next Oncology-Dallas, Irving, Texas
  - UT health east Texas HOPE Cancer Center, Tyler, Texas
  - Next Oncology-Virginia, Fairfax, Virginia
  - Summit Cancer Center, Spokane Valley, Washington
- China (6):
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jilin Provincial Cancer Hospital, Changchun, Jilin
  - The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang